CLINICAL TRIAL: NCT00478777
Title: A Multicenter, Single-Arm, Open-Label Expanded Access Program for Lenalidomide Plus Dexamethasone in Previously Treated Subjects With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Celgene (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MM-019; 2006-004532-73 (EudraCT Number)
Record Dates: First submitted 2007-05-23; First posted 2007-05-25 (Estimated); Results first posted 2011-11-03 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-09

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: CC-5013; Revlimid; Lenalidomide; Celgene; Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lenalidomide plus dexamethasone (Experimental): Lenalidomide administered orally, 25 mg daily (QD) for the first 21 days of each 28-day cycle. Pulse dexamethasone administered orally, 40 mg daily on Days 1-4, 9-12, and 17-20 for each 28-day cycle during Cycles 1 to 4 (approximately months 1-4). Beginning with Cycle 5 (approximately month 5), dexamethasone was to be reduced to 40 mg QD for Days 1-4 of each 28 day-cycle.
  Interventions: Drug: Lenalidomide; Drug: dexamethasone

INTERVENTIONS:
Drug: Lenalidomide — Oral lenalidomide at a dose of 25 mg daily for 21 days every 28 days. Treatment as tolerated until disease progression.
  Other Names: Revlimid®
Drug: dexamethasone — Oral pulse dexamethasone at a dose of 40 mg daily on days 1-4, 9-12, and 17-20 for each 28-day-cycle for cycles 1 through 4 (approximately months 1-4). Beginning cycle 5 (approximately month 5) dexamethasone is reduced to 40 mg daily for days 1-4 every 28 days.

SUMMARY:
This was a multicenter, open-label, single-arm phase 3B study of the combination lenalidomide plus pulse high-dose dexamethasone.

This study (CC-5013-MM-019) was set up and executed primarily as an expanded access program in Germany.

Screening procedures were to take place within 28 days prior to Cycle 1 Day 1 (baseline) with the exception of hematology assessments that were to be performed within 14 days prior to Cycle 1 Day 1. Randomization, blinding, and stratification were not applied in this open-label single-arm study.

Eligible subjects given open-label treatment and received treatment with lenalidomide plus high-dose dexamethasone in 28-day cycles.

Lenalidomide (hard capsules) was to be administered orally (PO) at a dose of 25 mg daily (QD) for the first 21 days of each 28-day cycle. According to the protocol, accrual of subjects to the study was to be terminated within 2 months of commercial availability of lenalidomide for this indication in Germany.

Upon discontinuation from study, minimal information was collected in order to identify when disease progressed.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form.
* Must be ≥18 years of age at the time of signing the informed consent form.
* Must be able to adhere to the study visit schedule and other protocol requirements.
* Must be diagnosed with multiple myeloma that is progressing after at least 2 cycles of anti-myeloma treatment or that has relapsed with progressive disease after treatment.
* Subjects may have been previously treated with thalidomide and/or radiation therapy. In addition, radiation therapy initiated prior to or at baseline (Day 1) may be given concurrently with study therapy, provided that all other eligibility criteria are satisfied.
* Subjects must discontinue all anti-myeloma drug or non-drug therapy prior to the first dose of study drug with the exception of radiation therapy initiated prior to or at baseline (Day 1).
* Measurable levels of myeloma paraprotein in serum (>0.5 g/dL) or urine (>0.2 g excreted in a 24-hour collection sample).
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
* Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; and 3) for at least 28 days after discontinuation from the study.

Exclusion Criteria:

* The presence of any of the following will exclude a subject from study enrollment:
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or lactating females.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Any of the following laboratory abnormalities:

  * Absolute neutrophil count (ANC) <1,000 cells/mm^3 (1.0 x 10^9/L)
  * Platelet count <75,000/mm^3 (75 x 109/L) for subjects in whom <50% of the bone marrow nucleated cells are plasma cells.
  * Platelet count <30,000/mm^3 (30x10^9/L) for subjects in whom ≥50% of bone marrow nucleated cells are plasma cells.
  * Serum creatinine >2.5 mg/dL (221 µmol/L)
  * Serum SGOT/AST or SGPT/ALT >3.0 x upper limit of normal (ULN)
  * Serum total bilirubin >2.0 mg/dL (34 µmol/L)
* Prior history of malignancies other than multiple myeloma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for ≥1 year.
* Prior history of stroke and/or thromboembolic event
* Known hypersensitivity to thalidomide or dexamethasone.
* Prior history of uncontrollable side effects to dexamethasone therapy.
* The development of a desquamating rash while taking thalidomide.
* Neuropathy ≥ Grade 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-03; Primary Completion 2007-11 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Axel Glasmacher, MD, Principal Investigator — University of Bonn
Locations (48):
- Germany (48):
  - Medizinische Klinik und Poliklinik II der Charité Universitätsmedizin Berlin Campus Mitte, Berlin
  - Poliklinik I, Hämatologie/ Onkologie, Universitätsklinikum Bonn, Bonn
  - Johanniter-Krankenhaus Bonn Friedrich-Wilhelm-Stift gGmbH, Bonn
  - Medizinische Klinik Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Interne Klinik Dr. Argirov, Schön-Kliniken, Burg
  - Klinik für Innere Medizin III Klinikum Chemnitz gGmbH, Chemnitz
  - Ärzte f. Innere Medizin Gemeinschaftspraxis f. Hämatologie u. Onkologie, Cologne
  - Klinik f. Innere Medizin, Klinikum der Universität zu Köln, Cologne
  - Medizinische Klinik und Poliklinik, Uniklinikum Dresden, Dresden
  - Universitaetsklinikum Dusseldorf Klinik fuer Haematologie, Düsseldorf
  - Direktor der Klinik f. Hämatologie, Universitätsklinikum Essen, Essen
  - Universitätsklinikum EssenInnere Klinik und Poliklinik, Essen
  - Klinik für Innere Medizin, Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder)
  - Medizinische Klinik II (ZIM),Hämatologie / Onkologie Uniklinik Frankfurt, Frankfurt am Main
  - Abt. Innere Medizin I , Hämatologie / Onkologie, Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum GöttingenHamatologie und Onkologie, Göttingen
  - Interdisziplinäre Klinik und Poliklinik für Stammzellentransplantation Universitätsklinik Hamburg - Eppendorf, Hamburg
  - II. Medizinische Abteilung, Asklepios Klinikum Altona, Hamburg
  - Abt. Hämatologie, Hämatologie und Onkologie, Medizinische Hochschule Hannover, Hanover
  - Medizinische Klinik und Poliklinik V Universitaetsklinikum Heidelberg, Heidelberg
  - Klinik für Innere Medizin II Hämatologie / Onkologie Universitätsklinikum Jena, Jena
  - EPS - Early Phase Solutions GmbH, Jena
  - Hämatologie / Onkologie / Infektionskrankheiten, Palliativmedizin Städtisches Klinikum Karlsruhe, Karlsruhe
  - 2. Med. Klinik , Sektion f. Stammzell- + Immuntherapie Universitätsklinikum Schleswig-Holstein, Kiel
  - Institut für Versorgungsforschung in der Onkologie Praxisklinik für Hämatologie und Onkologie, Koblenz
  - Medizinische Klinik und Poliklinik II Abt. Hämatologie / Onkologie, Universitätsklinikum Leipzig AÖR, Leipzig
  - III. Med. Klinik, Johannes Gutenberg Universität, Mainz
  - Klinikum Mannheim der Universität Heidelberg, Mannheim
  - Hämatologisch-Onkologisches Institut für medizinische Service Leistungen, Mönchengladbach
  - Medizinische Klinik III Klinikum der Universität München-Großhadern, München
  - Medizinische Klinik und Poliklinik A, Universitätsklinikum Münster, Münster
  - Fachärzte für Innere Medizin Hämatologie und Onkologie Gemeinschaftspraxis, Münster
  - Onkologie Praxis Oldenburg, Oldenburg
  - Abt. Onkologie/ Hämatologie, Klinikum Oldenburg, Oldenburg
  - Abteilung Hämatologie und Onkologie, Hämatologie und Onkologie, Medizinische Klinik, Klinikum Ernst v. Bergmann, Potsdam
  - Klinikum der Universität Regensburg, Regensburg
  - Abteilung Hämatologie und Onkologie, Medizinische Fakultät der Universität Rostock, Rostock
  - Caritasklinik St. Theresia, Saarbrücken
  - ms² Medizinische Statistik Saarbrücken, Saarbrücken
  - Med. Klinik III , St. Marienkrankenhaus Siegen, Siegen
  - Zentrum für Innere Medizin II Robert- Bosch-Krankenhaus GmBH, Stuttgart
  - Krankenanstalt Mutterhaus der Borromäerinnen, Trier
  - Abt. II Hämatologie, Onkologie und Immunologie Medizinische Klinik Abt.II, Tübingen
  - Medizinische Universitätsklinik, Ulm
  - Med. Klinik 1, Helios Klinikum Wuppertal, Wuppertal
  - Praxis Dres. Maintz & GroschekHämatologie / Onkologie, Würselen
  - Med. Klinik u. Poliklinik IIKlinikum der Universität Würzburg, Würzburg
  - Hämatologisch-onkologische Praxis, Würzburg

REFERENCES:
- [Result] Weisel, Katja Christina, et. al. Speed of Response with Lenalidomide and Dexamethasone in Patients with Relapsed or Refractory Multiple Myeloma: First Results of the MM-019 Compassionate Use Protocol. 14th Congress of the European Hematology Association, June 2009. Haematologica 2009; 94(Suppl 2):160 abs.0397. http://www.eventure-online.com/eventure/publicAbstractView.do?id=101710&congressId=2432

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 150 participants in 37 sites in Germany were enrolled when lenalidomide became commercially available in Germany. Study completion (end of study) was the time point when participants discontinued study drug and could switch to commercial lenalidomide.
Period: Overall Study
Arm/Group | Lenalidomide Plus Dexamethasone
Started | 150
Safety and Full Analysis Set (FAS) | 144 (6 enrolled participants did not receive lenalidomide.)
Completed | 73 (10 participants had >= 6 months and 63 participants < 6 months treatment prior to study termination.)
Not Completed | 77
Not completed — Adverse Event | 29
Not completed — Lack of Efficacy | 23
Not completed — Withdrawal by Subject | 4
Not completed — Death | 3
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 1
Not completed — Intolerance of therapy | 1
Not completed — Lack of compliance | 1
Not completed — Lymphocytes infusion | 1
Not completed — End of therapy | 2
Not completed — Not treated with lenalidomide | 6

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 144
Age Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 76
Race/Ethnicity, Customized [Number; unit: participants]
  White | 142
  Other | 2
Region of Enrollment [Number; unit: participants]
  Germany | 144

OUTCOME MEASURES:

1. Primary Outcome: Kaplan Meier Estimate for Time to Disease Progression
Description: Time to disease progression (TTP) was based on the European Group for Blood and Marrow Transplantation (EBMT) myeloma response determination criteria developed by Bladé (Bladé, 1998). TTP is a Kaplan Meier estimate of the time from randomization to the first documentation of progressive disease.
  Progressive disease based on increasing monoclonal paraprotein levels require a confirmatory value one week apart. Disease progression can also be based on bone marrow findings, worsening lytic bone disease, progressively enlarging extramedullary plasmacytomas, or hypercalcemia.
Time Frame: up to 827 days
Population: Full analysis dataset
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 144
days | 214.0 [146 to 281]

2. Secondary Outcome: Participant's Best Overall Response Based on the European Group for Blood and Marrow Transplantation (EBMT) Myeloma Response Criteria
Description: Best overall response was calculated as the best assessment from all cycles (including treatment discontinuation visit) and follow-up. The response rate was summarized as complete response (CR), partial response (PR), stable disease (SD), progression (PD), response not evaluable, and derived categories (PR+CR) and (PR+CR+SD).
  CR is negative immunofixation on both serum and urine maintained for 6 weeks straight. PR is a 50% decrease in serum paraprotein maintained for 6 weeks straight. SD is serum paraprotein values within 25% of baseline.
Time Frame: Up to 827 days
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 144
participants
  Complete response (CR) | 6
  Partial response (PR) | 97
  Stable disease (SD) | 30
  Progressive disease (PD) | 3
  Not evaluable (NE) | 8
  CR + PR | 103
  CR + PR + SD | 133

3. Secondary Outcome: Participants With Treatment-emergent Adverse Experiences (TEAEs)
Description: Counts of study participants who had treatment-emergent adverse events (TEAEs) defined as any reported AE that started on or after the first day of study drug dosing. A participant with multiple occurrences of an adverse event within a category is counted only once in that category.
  National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 3.0) was used by investigators to assess TEAEs. Severity scale ranges from 0 (none) to 5 (death). Grade 3=severe AE; Grade 4=life threatening or disabling AE; Grade 5=death.
Time Frame: up to 8 months
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 144
participants
  >=1 TEAE | 139
  >=1 TEAE related to study drug | 119
  >=1 NCI CTCAE grade 3 or 4 TEAE | 105
  >=1 NCI CTCAE grade 3 or 4 TEAE related to drug | 83
  >=1 serious AE (SAE) | 79
  >=1 study drug related SAE | 48
  Discontinued due to TEAE | 32
  Discontinued due to TEAE related to study drug | 21
  TEAE leading to dose reduction | 35
  TEAE leading to dose interruption | 64
  Deaths | 79

4. Secondary Outcome: Time to Partial Response Based on the European Group for Blood and Marrow Transplantation (EBMT) Myeloma Response Determination Criteria
Description: Time to partial response is the time from randomization to a 50% decrease in serum paraprotein maintained for six weeks straight. This was determined by free light chain concentrations which were taken every two weeks during the treatment phase of the trial.
Time Frame: up to 827 days
Population: Values for the free light chain concentrations were determined to be invalid.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 8 months
Arm/Group | Lenalidomide Plus Dexamethasone
Serious Adverse Events (participants affected / at risk) | 79/144
Other Adverse Events (participants affected / at risk) | 129/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide Plus Dexamethasone (N=144)
Pyrexia (General disorders) | 14
General physical health deterioration (General disorders) | 6
Asthenia (General disorders) | 2
Multi-organ failure (General disorders) | 2
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Gait disturbance (General disorders) | 1
Orthostatic intolerance (General disorders) | 1
Pain (General disorders) | 1
Pneumonia (Infections and infestations) | 8
Sepsis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Febrile infection (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 3
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Anal haemorrhage (Gastrointestinal disorders) | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Duodenitis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Large intestinal perforation (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Tooth disorder (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Grand mal convulsion (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Neurological symptom (Nervous system disorders) | 1
Neuromyopathy (Nervous system disorders) | 1
Syncope vasovagal (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 3
Atrial fibrillation (Cardiac disorders) | 2
Tachyarrhythmia (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Bundle branch block right (Cardiac disorders) | 1
Extrasystoles (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemia plasmacytic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal failure (Renal and urinary disorders) | 4
Renal failure acute (Renal and urinary disorders) | 3
Renal impairment (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis (Vascular disorders) | 3
Hypotension (Vascular disorders) | 2
Circulatory collapse (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Subclavian vein thrombosis (Vascular disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 1
Mental disorder due to a general medical condition (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Vertigo (Ear and labyrinth disorders) | 3
Haemoglobin decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Protein total increased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Epidermolysis bullosa (Congenital, familial and genetic disorders) | 1
Factor VIII deficiency (Congenital, familial and genetic disorders) | 1
Vision blurred (Eye disorders) | 1
Acute graft versus host disease in intestine (Immune system disorders) | 1
Graft versus host disease (Immune system disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide Plus Dexamethasone (N=144)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 35
Back pain (Musculoskeletal and connective tissue disorders) | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 8
Fatigue (General disorders) | 33
Oedema peripheral (General disorders) | 19
Pyrexia (General disorders) | 18
Dizziness (Nervous system disorders) | 17
Tremor (Nervous system disorders) | 15
Polyneuropathy (Nervous system disorders) | 14
Paraesthesia (Nervous system disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 22
Constipation (Gastrointestinal disorders) | 20
Nausea (Gastrointestinal disorders) | 9
Leukopenia (Blood and lymphatic system disorders) | 28
Thromboyctopenia (Blood and lymphatic system disorders) | 25
Anaemia (Blood and lymphatic system disorders) | 15
Lymphopenia (Blood and lymphatic system disorders) | 14
Neutropenia (Blood and lymphatic system disorders) | 12
Nasopharyngitis (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 9
Haemoglobin decreased (Investigations) | 13
C-reactive protein increased (Investigations) | 12
Insomnia (Psychiatric disorders) | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Multicenter publication must include input from investigators and Celgene, agreement to be established before publication. It has priority over subset (single center) publication, for duration of 1 year after study completion.
* Individual investigators have publication right after multicenter publication is complete (or 1 year after study completion), whichever is first. In this case, Celgene has the right to comment and right to ask delay of publication for 90 days.